CLINICAL TRIAL: NCT06829940
Title: Efficacy of Baduanjin Exercise in COVID-19 Contraction Patients With Idiopathic Chronic Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005517
Record Dates: First submitted 2025-02-14; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise training (Experimental): Each BET session consisted of a 10-minute warm-up and a 10-minute cool-down period [Xia et al., 2023]. These were followed by a 40-minute BET segment, which typically involved eight distinct body postures. These postures are based on the "Health Qigong Baduanjin Standard," as outlined in Zhao et al. [2019] and Koh [1982]. The eight postures are: (1) Support the Heaven, (2) Draw a Bow to Each Side, (3) Hold Up a Single Hand, (4) Practice Looking Back, (5) Shake the Hand and Wag the Tail, (6) Touch the Feet with Both Hands, (7) Climbing with Both Hands, and (8) Relax the Back, as explained in Zeng et al. [2020]
  Interventions: Other: Baduanjin exercise training (BET)
- waitlist (No Intervention): this group will receive no intervention

INTERVENTIONS:
Other: Baduanjin exercise training (BET) — Baduanjin Exercise Training (BET) is a traditional Chinese exercise focused on improving physical health, flexibility, balance, and mental well-being. It involves a 10-minute warm-up, a 40-minute core session practicing eight distinct postures, and a 10-minute cool-down. The postures, based on the Baduanjin form, target different body parts and promote strength, flexibility, and circulation. The exercises are synchronized with deep breathing to enhance relaxation and stress reduction. BET is especially beneficial for joint health, mobility, and mental clarity, making it suitable for individuals of all ages and fitness levels
  Arms: Baduanjin exercise training

SUMMARY:
Post-COVID recovery is associated with reduced functional fitness/capacity, low quality of life, and physical disabilities in those who survived after contracting the disease. The unpleasant symptoms of chronic post-viral/post-COVID syndrome (chronic fatigue perception, variant nonspecific myalgia, bad mood or depression, and insomnia or sleep disturbances) usually magnify the symptoms of already existing previously diagnosed concurrent untreatable chronic disorders , including the idiopathic chronic fatigue (ICF).(Leszczak et al., 2024)

Baduanjin exercise training (BET) is one of the Chinese traditional Health-Qigong exercises that not only integrate slow coordinating postures/positions, breathing techniques, musculoskeletal stretching movements/positions, and meditative mind but also plays a strong role concerning health benefits (e.g. musculoskeletal pain-reducing, sleep disturbance-enhancing effects, and fatigue-reducing effects) (Zou et al., 2018).

DETAILED DESCRIPTION:
forty idiopathic chronic fatigue (ICF) patients will be randomly assigned into two equal groups (n=20)

1. Study group (20 patients) this group will be supervised daily, except Fridays, during the 60-minute session of 12-week BET) or waitlist group
2. Control group (20 patients)

ELIGIBILITY:
Inclusion Criteria:

* • 40 patients will be recruited in the study.

  * age ≥ 18 to ≤ 50 years old
  * achieved three diagnostic items/criteria of ICF will be included in this BET trial: Fatigue lasting over 6 months, which significantly limits daily activities, reducing the person's usual activity level by more than 50%, as confirmed by a doctor.

At least three of the following symptoms:

Generalized muscle weakness Difficulty sleeping Frequent headaches A painful throat Muscle tenderness throughout the body Migratory joint pain Swollen lymph nodes in the neck or armpits Fatigue lasting more than a day after typical activities

Exclusion Criteria:

* Patients with a history of medical or complementary treatments for ICF disorder in the 6 months before contracting COVID or after recovery.
* Individuals who have engaged in therapeutic exercise, pharmacological treatments, or complementary therapies for post-COVID symptoms within the last six months prior to enrollment.
* ICF patients regularly using antidepressants or antipsychotics were excluded.
* Those who take sleeping pills regularly were also excluded.
* Patients with autoimmune diseases, malignant conditions, anemia, endocrine disorders, systemic diseases, or osteoarthritis affecting the cervical spine, lumbar region, or limbs were excluded.
* Individuals with abnormal results in laboratory tests, including neurological, neurophysiological, cardiological, liver/kidney function tests, or urine/stool analyses (as determined by a physician) were excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function: By Spirometry Device: | By Spirometry Device: forced vital capacity will be measured at baseline, and it will be measured after twelve weeks again
  • Pulmonary function: By Spirometry Device: it measure ventilatory functions. forced vital capacity (FVC)

SECONDARY OUTCOMES:
Pulmonary function: By Spirometry Device: | By Spirometry Device forced expiratory volume in one second (FEV1) will be measured at baseline, and it will be measured after twelve weeks again
  Pulmonary function: By Spirometry Device: it measure ventilatory functions forced expiratory volume in one second (FEV1)
Measuring functional capacity: By Six-minute walk test (6MWT) | Measuring functional capacity: By Six-minute walk test (6MWT)::will be measured at baseline, and it will be measured again after twelve weeks
  Measuring functional capacity: By Six-minute walk test (6MWT): is a self paced submaximal field exercise test , It will be performed according to the standard procedure is administered in a 30 meter hallway. (Launois et al., 2012 and ATS statement2002)
Modified Borg dyspnea scale (MBDS) | Modified Borg dyspnea scale (MBDS) will be measured at baseline, and it will be measured again after twelve weeks
  Modified Borg dyspnea scale (MBDS) is patient self-reported measures of one's difficulty in breathing upon exertion
Strength of lower limb muscles By a thirty-second sit-to-stand test | thirty-second sit-to-stand test will be measured at baseline, and it will be measured again after twelve weeks
  thirty-second sit-to-stand test was designed for testing leg strength and endurance it is the number of repetitions of sit-to-stand action executed in thirty seconds
Endurance of upper limb muscles: by the maximal repetitions of push-ups (MRPU). | the maximal repetitions of push-ups (MRPU). will be measured at baseline, and it will be measured again after twelve weeks
  Endurance of upper limb muscles: by the maximal repetitions of push-ups (MRPU) is commonly used to assess upper body strength, muscular endurance, and overall fitness levels.
Cardiorespiratory fitness:by the index of Ruffier test (IRT). | Cardiorespiratory fitness:by the index of Ruffier test (IRT). will be measured at baseline, and it will be measured again after twelve weeks
  Cardiorespiratory fitness: by the index of Ruffier test (IRT). is a simple, non-invasive method used to assess the recovery capacity of the heart after exercise and can be used to monitor fitness improvements over time.
Quality of life: by the short form 36 questionnaire (SF) | Quality of life: by the short form 36 questionnaire (SF) will be measured at baseline, and it will be measured again after twelve weeks
  Quality of life: by the short form 36 questionnaire (SF) is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used
sleep quality by Pittsburgh sleep quality index (PSQI): | sleep quality by Pittsburgh sleep quality index (PSQI):will be measured at baseline, and it will be measured again after twelve weeks
  sleep quality by Pittsburgh sleep quality index (PSQI): This is a 19 item widely used self-report questionnaire designed to assess sleep quality and disturbances
Beck Depression Inventory (BDI): | Beck Depression Inventory (BDI):will be measured at baseline, and it will be measured again after twelve weeks
  Beck Depression Inventory (BDI):widely used self-report questionnaire designed to assess the presence and severity of depressive symptoms
fatigue assessment by Buzhongyiqi-Tang questionnaire (BZTQ): | Buzhongyiqi-Tang questionnaire (BZTQ)::will be measured at baseline, and it will be measured again after twelve weeks
  Buzhongyiqi-Tang questionnaire (BZTQ): Fatigue syndrome's severity can be rated via this validated 16-item questionnaire (every item was rated 7-Likert scale responses starting from zero to seven).

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-moatasem, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt